CLINICAL TRIAL: NCT00834353
Title: Prospective Study of N-acetyltransferase2 (NAT2) Gene and Rifampicin Induced Cytochrome P-450 as Susceptible Risk Factors for Antituberculosis Drug Induced Hepatitis
Brief Title: Prospective Study of N-acetyltransferase2 (NAT2) and Cytochrome P4502E1 (CYP2E1) Gene as Susceptible Risk Factors for Antituberculosis (ATT) Induced Hepatitis
Status: Completed | Type: Observational
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Dr. Premashis kar, Director Professor, Deptt. Medicine, MAMC, New Delhi
Other Study IDs: F.501(134)/02-EC/MC(Aca)/16713
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmonary tuberculosis patients: Freshly diagnosed pulmonary tuberculosis patients who are started with antituberculosis drugs
  Interventions: Drug: ATT

INTERVENTIONS:
Drug: ATT

SUMMARY:
N-acetyltransferase2 (NAT2) and Cytochrome P4502E1 (CYP2E1) are two drug metabolizing enzymes. Antituberculosis drug isoniazid is acetylated by NAT2 and forms ultimately a nontoxic compound which is metabolized by CYP2E1 to a toxic metabolite. Slow acetylator genotype of NAT2 and wild type genotype of CYP2E1 gene has been attributed to greater toxicity of ATT drug. Therefore this study has been designed to analyze the genetic polymorphism of NAT2 and CYP2E1 genes in tuberculosis patients who developed drug induced hepatitis upon administration of antituberculosis drug.Polymorphism study of NAT2 and CYP2E1 gene may help in predicting the high risk group of ATT induced hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary tuberculosis
* Patients receiving conventional antituberculosis drugs
* Patients who directly presented with antituberculosis drug induced hepatitis

Exclusion Criteria:

* Habitual alcohol drinkers
* Patients with evidence of viral hepatitis

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases are enrolled in the study from primary care clinic after they are diagnosed with pulmonary tuberculosis.
Sampling Method: Probability Sample
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premashis Kar, MD,DM, Principal Investigator — Maulana Azad Medical College, Department of Medicine.
Locations (1):
- Premashis Kar, New Delhi, New Delhi, India